CLINICAL TRIAL: NCT07318532
Title: Socio-Structural Intervention to Improve Pre-Exposure Prophylaxis (PrEP) Services for Cisgender Women (CGW) (PrEP-CGW)
Brief Title: Socio-Structural Intervention to Improve Pre-Exposure Prophylaxis Services for Cisgender Women
Acronym: PrEP CGW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: MedstarRI; R34MH128046 (NIH)
Record Dates: First submitted 2026-01-02; First posted 2026-01-06 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2025-12

CONDITIONS: HIV Prevention Program
Keywords: HIV pre-exposure prophylaxis (PrEP); HIV prevention; Women

STUDY DESIGN:
Intervention Model Description: Note, this is a clinic-level intervention. Thus the "participant" is the clinic.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PrEP CGW Pilot: W-PrEP intervention arm (Experimental): W-PrEP intervention arm included exposure to trained providers and clinic staff, PrEP navigation, and patient-facing educational resources such as videos, pamphlets, posters, and an educational website.
  This arm was compared to historical controls from the same calendar year.
  Interventions: Behavioral: The women's PrEP Project (W-PrEP)

INTERVENTIONS:
Behavioral: The women's PrEP Project (W-PrEP) — W-PrEP intervention included exposure to trained providers and clinic staff, PrEP navigation, and patient-facing educational resources such as videos, pamphlets, posters, and an educational website.
  Other Names: W-PrEP

SUMMARY:
The goal of the "PrEP CGW" pilot study is evaluate the feasibility and acceptability of a clinic-level intervention to improve HIV prevention and Pre-exposure Prophylaxis (PrEP) services for women. The intervention includes clinic wide trainings, provider and clinic staff tool kits, PrEP navigation, and patient-facing educational resources. The overarching goal of the program is to determine if the intervention improves PrEP uptake among women.

Patients who attend the study-site clinic will be exposed to the intervention. Patients will be invited to participate in post-visit questionnaires; approximately 20 patients will be invited to participate in interviews.

DETAILED DESCRIPTION:
The goal of the "PrEP CGW" pilot study is evaluate the feasibility and acceptability of a clinic-level intervention to improve HIV prevention and Pre-exposure Prophylaxis (PrEP) services for women. Feasibility testing additionally includes assessing the appropriateness of the study measures (e.g., questionnaires, interviews, collection of electronic health record data) to assess the outcomes of interest in the planned full scale trial. The intervention includes clinic wide trainings, provider and clinic staff tool kits, PrEP navigation, and patient-facing educational resources developed and/or collated as part of the R34 award. The overarching goal of the program is to determine if the intervention improves PrEP uptake among women.

Patients who attend the study-site clinic will be exposed to the clinic level intervention. Patients will be invited to participate in post-visit questionnaires; approximately 20 patients will be invited to participate in interviews. Electronic health data from the intervention period will be compared with a historical control period.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care at the study-site clinic

Exclusion Criteria:

* N/A

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Cisgender women
Enrollment: 745 (Actual)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-04-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Reach | Each study visit within the 4 month intervention period
  * Percentage of eligible patients who received introduction to pre-exposure prophylaxis (PrEP) by navigators (by comparison of the navigators counseling log to the electronic health record (EHR)
  * Percentage of eligible patients counseled about PrEP by providers (by EHR review)
  * Percentage of eligible patients counseled by either the PrEP navigator or a provider

SECONDARY OUTCOMES:
Adoption | Two-month intervention training period
  * Percentage of clinic-team members who participated in training (by attendance log)
  * Percentage of change in PrEP knowledge and PrEP best practices (pre-/post-clinic-wide training questionnaire)
Intervention characteristics: organizational and patient perspectives | 6 months (four month intervention and two months of follow-up)
  * Perceived feasibility of implementing the intervention and identified barriers (by in depth interviews (IDI) with the clinic team and navigators)
  * Satisfaction with training and intervention usability/complexity among clinic team and navigators (by IDIs with the clinic team and navigators)
  * Acceptability of the provider or navigator PrEP education/counseling, focusing on burden and addressing patient barriers (by IDI with patients)

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Scott R, Hull SJ, Kerrigan D, Wang Y, Pratt-Chapman M, Mathias-Prabhu T, Unwala N, Sadauskas M, Hose BZ, Smith M, Moriarty P, Hanson T, Tedla A, Lotke P, Ye P, Arem H. "The Women's PrEP Project," a Clinic-Based, Socio-Structural Intervention to Improve the Provision of Preexposure Prophylaxis for Cisgender Women: Interrupted Time Series Pilot. JMIR Form Res. 2025 Dec 3;9:e80653. doi: 10.2196/80653. PMID 41337677

DOCUMENTS (1):
  • Statistical Analysis Plan (2021-05-03): https://cdn.clinicaltrials.gov/large-docs/32/NCT07318532/SAP_000.pdf